CLINICAL TRIAL: NCT01724749
Title: Cardiovascular Molecular Calcification Assessed by 18F-NaF PET CT: The CAMONA Study
Brief Title: Cardiovascular Molecular Calcification Assessed by 18F-NaF PET CT
Acronym: CAMONA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Björn A Blomberg, MD, MSc, Odense University Hospital
Other Study IDs: s-20120056
Record Dates: First submitted 2012-11-06; First posted 2012-11-12 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Cardiovascular Disease; Atherosclerosis; Angina Pectoris
Keywords: Atherosclerosis; Sodium-Fluoride; 18F-Sodium Fluoride; 18F-NaF; fluorodeoxyglucose; 18F-FDG; FDG; Positron emission tomography; PET
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy control subjects: 1. Age: 21 - 80 years
  2. No prior history or symptoms of cardiovascular disease
  The investigators aim to include equal numbers of females and males. Furthermore, the investigators aim to include patients in six different age strata: 21-30, 31-40, 41-50, 51-60, 61-70, 71-80.
- Subjects with cardiovascular disease: 1. Age: 21 - 80 years
  2. HeartSCORE > 0%
  3. Symptoms of angina pectoris
  The investigators aim to include equal numbers of females and males. Furthermore, the investigators aim to include patients in six different age strata: 21-30, 31-40, 41-50, 51-60, 61-70, 71-80. Also, the investigators aim to include patients in 3 strata of HeartSCORE risk: low risk (1-4%), mild risk (5-9%) and high risk (> 9%)

SUMMARY:
The purpose of the CAMONA study is to demonstrate the feasibility of cardiovascular molecular calcification (CMC) assessment by means of 18F-sodium-fluoride (18F-NaF) positron emission tomography (PET) computed tomography (CT) in a prospective cohort of healthy control subjects and subjects with cardiovascular disease.

DETAILED DESCRIPTION:
Atherosclerosis associated cardiovascular disease (CVD) remains a significant cause of morbidity and mortality. Asymptomatic individuals with a moderate to high-risk of developing acute atherosclerotic cardiovascular events will benefit most from intensive evidence-based medical interventions.

The traditional approach to identify patients with moderate to high-risk of CVD involves quantifying the presence of CVD risk factors. Based on gender, age, smoking, systolic blood pressure and cholesterol levels, risk stratification algorithms such as the Framingham Risk Score (FRS) and the European SCORE system can predict the 10-year risk of cardiovascular death.

However, these algorithms are associated with several limitations, including misclassification of women and individuals with high levels of a single risk factor. The risk is underestimated in these individuals. Therefore, these individuals are not eligible for treatment by current criteria of CVD prevention guidelines. Several studies indicate that the traditional risk score models leave room for improvement, as they work reasonably well for populations, but remain suboptimal for individual subjects.

New risk parameters are discovered on a regular basis. One of these parameters is cardiovascular molecular calcification (CMC). This entity can be detected and quantified by 18F-NaF PET CT. It has been hypothesized that CMC can be detected years, maybe even decades, before coronary artery calcium scoring (CACS) can be detected by conventional imaging modalities like multislice CT. Theoretically, this tool can detect patients at a very early stage of the disease. Providing evidence-based treatment to these individuals can, theoretically, improve the prevention of CVD. Before this hypothesises can be tested, the feasibility of 18F-NaF PET CT has to be demonstrated in both healthy controls as well as in subjects with cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21 - 80 years
* Healthy controls: No prior history or symptoms of cardiovascular disease
* Cardiology subjects: Eligibility for CACS due to symptoms suggesting angina pectoris.
* Cardiology subjects: HeartSCORE > 0%.

Exclusion Criteria:

* Pregnancy
* Extensive physical activity or extensive partying passed 24 hours
* History of malignant neoplasms with past 5 years
* Known immunodeficiencies
* History of deep vein thrombosis or acute pulmonary embolism within the previous three months
* History of alcohol abuses, illicit drug use, or drug abuse, or significant mental illness
* Initiation of statin-therapy within 3 months prior to consideration of study enrolment
* History of autoimmune disease, such as systemic lupus erythematosus, inflammatory bowel disease, sarcoidosis, rheumatoid arthritis, or psoriasis.
* Participation in any clinical trial of an investigational drug, device, or medical procedure within 30 days prior to baseline of the study
* Enrolment or planned enrolment in another clinical trial during the study period

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy control subjects will be recruited from a random sample of Danish citizens. To secure timely inclusion of healthy controls, blood donors will be approached for inclusion as well.
  Subjects with symptoms suggesting angina pectoris will be recruited from the Department of Cardiology, Odense University Hospital. Each patient referred for symptoms suggesting angina pectoris and eligibility for a coronary artery calcium scoring (CACS) will be eligible for inclusion in the investigators study.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) of 18F-NaF | Up to 7 days after the day of PET CT acquisition
  The SUV is a validated semi-quantitative assessment of PET radiotracer uptake. The SUV of 18F-NaF will be determined in the aorta, carotid arteries, coronary arteries, iliac arteries and the femoral arteries.
Target to background ratio (TBR) of 18F-NaF | Up to 7 days after the day of PET CT acquisition
  The TBR is a validated semi-quantitative assessment of PET radiotracer uptake. The TBR of 18F-NaF will be determined in the aorta, carotid arteries, coronary arteries, iliac arteries and the femoral arteries.

SECONDARY OUTCOMES:
Standardized uptake value (SUV) of 18F-Fluorodeoxyglucose (18F-FDG) | Up to 7 days after the day of PET CT acquisition
  The SUV is a validated semi-quantitative assessment of PET radiotracer uptake. The SUV of 18F-FDG will be determined in the aorta, carotid arteries, iliac arteries and the femoral arteries.
Target to background ratio (TBR) of 18F-FDG | Up to 7 days after the day of PET CT acquisition
  The TBR is a validated semi-quantitative assessment of PET radiotracer uptake. The TBR of 18F-FDG will be determined in the aorta, carotid arteries, iliac arteries and the femoral arteries.
Correlation between the TBR of 18F-NaF/18F-FDG and traditional cardiovascular risk factors. | The cardiovascular risk factors will be determined, on average, 1 hour before 18F-NaF / 18F-FDG injection; which ever comes first
  The traditional cardiovascular risk factors consist of:
  1. Smoking, pack years;
  2. Alcohol, units/week;
  3. Blood pressure, mean arterial pressure, mmHg;
  4. Body mass index, kg/m2;
  5. Waist circumference, cm;
  6. History of cardiovascular disease;
  7. Family history of cardiovascular disease;
  8. Medication usage;
  9. Age;
  10. Gender.
Correlation between the TBR of 18F-NaF/18F-FDG and blood markers of atherosclerosis. | The blood draw will be performed, on average, 1 hour before the 18F-FDG PET CT scan and the blood markers will determined in upto 48 hours after the 18F-FDG PET CT scan
  Blood markers:
  1. Total cholesterol, mmol/L;
  2. LDL cholesterol, mmol/L;
  3. HDL cholesterol, mmol/L;
  4. Triglycerides, mmol/L;
  5. Homocysteine, mmol/L;
  6. Fasting plasma glucose, mmol/L;
  7. HBA1c, mmol/mol;
  8. High sensitivity C-reactive protein, nmol/L;
  9. Fibrinogen, umol/L;
  10. Leukocyte differentiation, cells/L;
  11. Creatinine, umol/L;
Correlations between 18F-NaF TBR, 18F-FDG TBR, and CT calcification scoring | Up to 7 days after the day of PET CT acquisition
  Correlation between the degree of 18F-NaF uptake, 18F-FDG uptake, CT-Calcification scoring and the various arterial segments (aorta, carotid arteries, iliac arteries and the femoral arteries.
Target to background ratio (TBR) of 18F-NaF | Up to 7 days after the day of PET CT acquisition
  18F-NaF PET/CT images will be acquired at 45, 90 and 180 minutes after intravenous injection of the compound in a subset of 40 patients. The TBR of 18F-NaF will be determined at each time point and compared to allow determining the optimum tracer circulation time for maximum contrast between the vessel wall and blood pool.
Target to background ratio (TBR) of 18F-FDG | Up to 7 days after the day of PET CT acquisition
  18F-FDG PET/CT images will be acquired at 90 and 180 minutes after intravenous injection of the compound in a subset of 40 patients. The TBR of 18F-NaF will be determined at both time points and compared to allow determining the optimum tracer circulation time for maximum contrast between the vessel wall and blood pool.
Correlation between 18F-NaF / 18F-FDG uptake and 18F-FDG uptake in the brain | Up to 7 days after the day of PET CT acquisition
  18F-FDG uptake in the brain will be quantified by calculating the mean and maximum partial-volume corrected SUV.
Correlation between 18F-NaF TBR and 18F-NaF TBR two years after the baseline scan. | 2 years
  The TBR will be determined in various segments of the arterial tree.
Correlation between 18F-FDG TBR and 18F-FDG TBR two years after the baseline scan. | 2 years
  The TBR will be determined in various segments of the arterial tree.
Correlation between the TBR of 18F-NaF/18F-FDG and HeartSCORE | Up to 7 days after the day of PET CT acquisition
  The HeartSCORE will be calculated according to the current HeartSCORE protocol for Denmark.
Correlation between the TBR of 18F-NaF/18F-FDG and Framingham Risk Score | Up to 7 days after the day of PET CT acquisition
  The Framingham Risk Score will be calculated according to the current recommendations by the Framingham Heart Study group
Correlation between 18F-NaF / 18F-FDG uptake and 18F-NaF / 18F-FDG uptake in the vertebral body | Up to 7 days after the day of PET CT acquisition
  18F-NaF uptake in the 1st, 3rd and 5th lumbar vertebral body will be quantified by calculating the mean and maximum partial-volume corrected SUV.
Arterial Calcification Score | Up to 7 days after the day of PET CT acquisition
  Arterial Calcification Scoring will be determined in Agatston Units as well as in volumetric units in all segments of the arterial tree (coronary arteries, aorta, carotid arteries, iliac and femoral arteries.

CONTACTS AND LOCATIONS:
Overall Officials: Poul F Høilund-Carlsen, MD, DMSc, Study Chair — Odense University Hospital; Björn A Blomberg, MD, MSc, Principal Investigator — Odense University Hospital
Locations (2):
- Denmark (2):
  - Department of Cardiology, Odense University Hospital, Odense, Region Syddanmark
  - Department of Nuclear Medicine, Odense University Hospital, Odense, Region Syddanmark

REFERENCES:
- [Derived] Patil S, Kata R, Teichner E, Subtirelu R, Ghonim M, Ghonim M, Al-Daoud O, Ismoilov M, Herpin L, Ayubcha C, Werner T, Hoilund-Carlsen PF, Alavi A. Associations of subclinical microcalcification and inflammation with carotid atheroma development: a dual-tracer PET/CT study. Eur J Nucl Med Mol Imaging. 2025 Jun;52(7):2502-2512. doi: 10.1007/s00259-025-07127-z. Epub 2025 Feb 13. PMID 39939531
- [Derived] Sorci O, Batzdorf AS, Mayer M, Rhodes S, Peng M, Jankelovits AR, Hornyak JN, Gerke O, Hoilund-Carlsen PF, Alavi A, Rajapakse CS. 18F-sodium fluoride PET/CT provides prognostic clarity compared to calcium and Framingham risk scoring when addressing whole-heart arterial calcification. Eur J Nucl Med Mol Imaging. 2020 Jul;47(7):1678-1687. doi: 10.1007/s00259-019-04590-3. Epub 2019 Nov 16. PMID 31734781
- [Derived] Pourhassan Shamchi S, Khosravi M, Taghvaei R, Zirakchian Zadeh M, Paydary K, Emamzadehfard S, Werner TJ, Hoilund-Carlsen PF, Alavi A. Normal patterns of regional brain 18F-FDG uptake in normal aging. Hell J Nucl Med. 2018 Sep-Dec;21(3):175-180. doi: 10.1967/s002449910902. Epub 2018 Nov 10. PMID 30411727